CLINICAL TRIAL: NCT02289638
Title: First Comparison of the /Intubrite VideoLaryngoscope System Versus the Miller Laryngoscope for Intubations by Non-anaesthetists: a Manikin Study.
Brief Title: Effectiveness of Child Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Institute of Cardiology, Warsaw, Poland, International Institute of Rescue Research and Education
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/13
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
Keywords: intubation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation without chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation without chest compressions.
  Interventions: Device: Intubrite; Device: MIL
- Intubation with uninterrupted chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: Intubrite; Device: MIL

INTERVENTIONS:
Device: Intubrite — Video-Laryngoscopy
  Other Names: Intubrite Video Laryngoscope System VLS 6600
Device: MIL — Direct-Laryngoscopy
  Other Names: Miller Laryngoscope

SUMMARY:
We hypothesized that the Intubrite Video Laryngoscope System VLS 6600 is beneficial for intubation of pediatric manikins while performing CPR. In the current study, we compared effectiveness of the Intubrite and MIL laryngoscopes in child resuscitation with and without CC.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (physicians, nurses, paramedics)

Exclusion Criteria:

* Not meet the above criteria
* Wrist or Low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of first, second and third intubation attempts and overall effectiveness of intubation by participants

SECONDARY OUTCOMES:
Intubation time | 1 day
  time in seconds required for a successful intubation attempt
POGO score | 1 day
  self-reported percentage of glottis opening (POGO) score
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland